CLINICAL TRIAL: NCT00260793
Title: Open Label Prospective Study of High Dose Ropinirole for Motor Fluctuations and Dyskinesias in Advanced Parkinson's Disease
Brief Title: Open Label High Dose Ropinirole (Requip) Study for Patients With Parkinson's Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Agarwal, Pinky, M.D. (Individual)
Collaborators: Colorado Neurology (Other); GlaxoSmithKline (Industry)
Organization: Colorado Neurology (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 103911
Record Dates: First submitted 2005-12-01; First posted 2005-12-02 (Estimated); Last update posted 2006-02-03 (Estimated); Status verified 2005-11

CONDITIONS: Parkinson's Disease
Keywords: Ropinirole; Parkinson's disease; dopamine agonist
MeSH Terms: conditions — Parkinson Disease | interventions — ropinirole

INTERVENTIONS:
Drug: Ropinirole Hydrochloride

SUMMARY:
The purpose of this research study is to see if subjects with Parkinson's disease who are experiencing motor fluctuations ("on" and "off" states) and dyskinesias (involuntary excessive movements) would benefit from a higher dose of Requip as compared to the maximum FDA approved dose of dopamine agonist drugs (including Requip, Mirapex, and Permax). Requip as used in this study is investigational, which means it has not been approved by the US Food and Drug Administration (FDA) at this dose level.

ELIGIBILITY:
Inclusion Criteria:

* Patients must give written informed consent prior to any specific study procedures.
* Males or females; females of childbearing age who are not currently pregnant must agree to use a medically accepted method of contraception throughout the study.
* Age greater than or equal to 25 years.
* Patients must be on a maximum dose of dopamine agonist drug (pergolide 4mg/day, pramipexole 4.5 mg/day or ropinirole 24mg/day).
* Stable dose of all medications for 4 weeks.

Exclusion Criteria:

* Current hallucinations.
* History of disabling hallucinations or hallucinations in past requiring treatment.
* Troublesome edema (swelling).
* Unstable depression.
* Female who is pregnant or lactating.
* Use of an investigational drug with in the last 30 days.
* Other inclusion or exclusion criteria to be evaluated by the physician.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-11

CONTACTS AND LOCATIONS:
Overall Officials: Pinky Agarwal, MD, Principal Investigator — Colorado Neurology, P.C.
Locations (1):
- Colorado Neurology, P.C., Englewood, Colorado, United States